CLINICAL TRIAL: NCT01791491
Title: A Phase 2 Multi-Center, Randomized Conversion Study to Evaluate the Pharmacokinetics, Efficacy, and Safety of Belatacept Administered to Pediatric Subjects With a Stable Renal Transplant
Brief Title: Pharmacokinetics, Safety and Tolerability of Single-dose Belatacept in Adolescent Kidney Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM103-144; 2011-005257-31 (EudraCT Number)
Record Dates: First submitted 2013-01-31; First posted 2013-02-15 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belatacept (Experimental)
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Belatacept — Single intravenous infusion of belatacept, 7.5 mg/kg
  Other Names: BMS-224818

SUMMARY:
The purpose of this study is to evaluate how well adolescent kidney transplant patients tolerate a single dose of belatacept they receive at least 6 months after transplant surgery, and how their body handles the drug.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male and Female subjects,12-17 years old
* Receiving CNI-based maintenance immunosuppression since the time of renal transplantation in accordance with local standard of care
* Stable renal function, in the opinion of the investigator, with a cGFR>45 mL/min/1.73m2 at the time of enrollment (per updated Schwartz Formula)
* Adolescent Recipients of a renal allograft from a living donor or a deceased donor at least 6 months prior to enrollment
* Subject must be receiving a calcineurin inhibitor (CNI)-based [cyclosporine (CsA) [any formulation] or Tacrolimus (TAC)] immunosuppressive regimen
* Subject must be receiving adjunctive background maintenance immunosuppression with mycophenolate mofetil (MMF) or enteric-coated mycophenolate sodium (EC-MPS)/mycophenolic acid (MPA)
* Subjects may be receiving maintenance corticosteroids in accordance with the local standard of care
* Negative Interferon Gamma Release Assay (IGRA) such as QuantiFERON-TB Gold test or T-Spot-TB
* FOCBP must have negative serum or urine pregnancy test within 24 hrs prior to start of study medication
* Subject must have stable estimated glomerular filtration rate (GFR) ≥45 mL/min/1.73m2 (updated Schwartz formula)

Exclusion Criteria:

* Epstein-Barr virus (EBV) serostatus negative or unknown at time of transplant and screening
* History of any treated or biopsy proven acute rejection (BPAR) within 3 months prior to enrollment
* Subjects who have experienced more than 1 episode of acute rejection (AR) of the current allograft or any antibody-mediated AR
* Subjects with any active infection [including, but not limited to, positive cytomegalovirus (CMV) or BK viral (BKV) loads, BKV associated nephropathy (BKVAN), CMV retinitis, CMV colitis, etc.]
* Urine albumin:creatinine ratio > 56.5 mg/mmol (> 0.5 mg albumin / mg creatinine) on a random voided urine specimen

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2013-05-09 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (8):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Childrens Hospital Of La, Los Angeles, California
  - University Of California Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Boston Childrens Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 participants were enrolled and 9 were treated. Reasons for non-treatment: 1 withdrew consent and 6 no longer met study criteria.
Groups:
- Belatacept: A single dose of 7.5 mg/kg Belatacept was given intravenously on study Day 1 over approximately 30 minutes.
Period: Overall Study
Arm/Group | Belatacept
Started | 9 (Reasons for enrollment and non-treatment: 1 withdrew consent and 6 no longer met study criteria.)
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Belatacept
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (1.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), and Treatment-related Adverse Event (AE)
Description: Death was a fatal event leading to permanent cessations of all vital functions of the body. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Adverse event (AE) defined: any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Treatment related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: Date of First Dose to 24 weeks post the last dose; approximately 26 weeks
Population: All treated participants who received at least one dose of belatacept.
Measure: Number; unit: participants
Arm/Group | Belatacept
Number analyzed (Participants) | 9
participants
  Death | 0
  SAEs | 4
  Treatment-related AEs | 0

2. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Belatacept
Description: Cmax was derived from serum concentration versus time data. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: pre-dose (0 hours), 0.5 and 2 hours from Start of Infusion on Day 1, Day 29, and Day 57. The results were summarized. The lower limit of assay quantitation (LLOQ) was set to "zero" which was 0.003 micrograms per milliliter (ug/mL). Cmax was measured in micrograms per milliliter.
Time Frame: Pre-dose (0), 0.5hr and 2hr from the start of infusion on Day 1, Day 29, and Day 57
Population: Pharmacokinetic (PK) analysis set: all participants who received one dose of belatacept and who had at least 1 blood sample drawn for PK determination.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | Belatacept
Number analyzed (Participants) | 9
micrograms per milliliter | 151 (20)

3. Primary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of Belatacept
Description: Tmax was derived from serum concentration versus time data. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: pre-dose (0 hours), 0.5 and 2 hours from Start of Infusion on Day 1, Day 29, and Day 57. The results were summarized. The lower limit of assay quantitation (LLOQ) was set to "zero" which was 0.003 micrograms per milliliter (ug/mL). Tmax was measured in hours (h).
Time Frame: Pre-dose (0), 0.5hr and 2hr from the start of infusion on Day 1, Day 29, and Day 57
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Belatacept
Number analyzed (Participants) | 9
hours | 0.733 [0.450 to 2.05]

4. Primary Outcome: Half-Life of Elimination (T-Half) of Belatacept
Description: T-HALF was derived from serum concentration versus time data. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: pre-dose (0 hours), 0.5 and 2 hours from Start of Infusion on Day 1, Day 29, and Day 57. The results were summarized. The lower limit of assay quantitation (LLOQ) was set to "zero" which was 0.003 micrograms per milliliter (ug/mL). T-HALF was measured in hours (h).
Time Frame: Pre-dose (0), 0.5hr and 2hr from the start of infusion on Day 1, Day 29, and Day 57
Population: Pharmacokinetic (PK) analysis set: all participants who received one dose of belataceptand who had at least 1 blood sample drawn for PK determination.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Belatacept
Number analyzed (Participants) | 9
hours | 173 (46.8)

5. Primary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC (0-T)) and Area Under the Serum Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC(INF)) of Belatacept
Description: AUC (0 - T) and AUC (0 - INF) were derived from serum concentration versus time data and measured in microgram hours per milliliter (µg*h/mL). Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: pre-dose (0 hours), 0.5 and 2 hours from Start of Infusion on Day 1, Day 29, and Day 57. The results were summarized. The lower limit of assay quantitation (LLOQ) was set to "zero" which was 0.003 micrograms per milliliter (ug/mL).
Time Frame: Pre-dose (0), 0.5hr and 2hr from the start of infusion on Day 1, Day 29, and Day 57
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram hours per milliliter
Arm/Group | Belatacept
Number analyzed (Participants) | 9
microgram hours per milliliter
  AUC (0-T) | 15145 (25)
  AUC(INF) | 15407 (25)

6. Primary Outcome: Total Body Clearance (CLT) of Belatacept
Description: CLT was the volume of abatacept cleared by the system, normalized by baseline body weight. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: pre-dose (0 hours), 0.5 and 2 hours from Start of Infusion on Day 1, Day 29, and Day 57. The results were summarized. The lower limit of assay quantitation (LLOQ) was set to "zero" which was 0.003 micrograms per milliliter (ug/mL). CLT was measured in milliliters per hours per kilogram of body weight (mL/h/kg).
Time Frame: Pre-dose (0), 0.5hr and 2hr from the start of infusion on Day 1, Day 29, and Day 57
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per hours per kilogram
Arm/Group | Belatacept
Number analyzed (Participants) | 9
milliliters per hours per kilogram | 0.483 (27)

7. Primary Outcome: Volume of Distribution at Steady-state (Vss) of Belatacept
Description: Vss was derived from serum concentration versus time data. Serum samples were analyzed for abatacept by a validated enzyme-linked immunosorbent assay (ELISA) and were obtained at: pre-dose (0 hours), 0.5 and 2 hours from Start of Infusion on Day 1, Day 29, and Day 57. The results were summarized. The lower limit of assay quantitation (LLOQ) was set to "zero" which was 0.003 micrograms per milliliter (ug/mL). Vss was measured in liters per kg body weight (L/kg).
Time Frame: Pre-dose (0), 0.5hr and 2hr from the start of infusion on Day 1, Day 29, and Day 57
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per kilogram
Arm/Group | Belatacept
Number analyzed (Participants) | 9
Liters per kilogram | 0.088 (30)

8. Secondary Outcome: Number of Participants With Positive Belatacept-induced Immunogenicity Response
Description: Serum samples were analyzed for anti-belatacept antibodies using a validated homogenous bridging assay. The assay followed a tiered approach consistent with health authority guidance: tier 1 for screening ADA responses, tier 2 for confirming drug specificity of the ADA-positive responses, and tier 3 for titer. A neutralizing antibody assay was used to test those samples positive to the LEA29Y portion of the molecule in tier 2 and for which drug concentrations are =>1 μg/mL. Lack of immunogenicity was defined as the absence of a positive response.
Time Frame: Baseline/Day 1, Days 15, 29, and 57
Population: All treated participants who received at least one dose of belatacept.
Measure: Number; unit: participants
Arm/Group | Belatacept
Number analyzed (Participants) | 9
participants | 0

9. Secondary Outcome: Percentage of CD86 Receptor Occupancy
Description: Blood samples collected following the single dose belatacept infusion were assessed for CD86 receptor occupancy (CD86 RO).
Time Frame: 0.5 hours post dose on Day 1, Day 29 and Day 57
Population: Pharmacodynamic analysis set: all participants who received one dose of belatacept and who had at least 1 pharmacodynamic result (CD86 RO) reported after that dose.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Belatacept
Number analyzed (Participants) | 7
percent
  0.5 Hour | 94.70 (4.035)
  Day 29 | 77.99 (10.983)
  Day 57: number analyzed (Participants) | 5
  Day 57 | 51.45 (43.285)

ADVERSE EVENTS:
Time Frame: SAEs were reported from the date of first dose to 24 weeks post the last dose (approximately 26 weeks); AEs were reported for the on study period from the date of first dose up to 56 days post last dose (approximately 10 weeks)
Arm/Group | Belatacept
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belatacept (N=9)
Gastroenteritis (Infections and infestations) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belatacept (N=9)
Headache (Nervous system disorders) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Asthenia (General disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.